CLINICAL TRIAL: NCT02621567
Title: Bright Light Therapy Efficacy for Depressive Symptoms Following Cardiac Surgery or Acute Coronary Syndrome: Pilot Trial
Acronym: BEAM-P
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Mark Eisenberg, Professor of Medicine, McGill University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-125
Record Dates: First submitted 2015-11-27; First posted 2015-12-03 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Depressive Symptoms Post Cardiac Surgery or Post Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bright Light Therapy Group (Experimental): Participants in this group will receive bright light therapy lamps and will be instructed to use them for 30 minutes every morning within an hour of waking up, everyday for 4 weeks.
  Interventions: Device: Bright Light Therapy Lamp
- Dim Light Group (Placebo Comparator): Participants in this group will receive modified dim lamps and will be instructed to use them for 30 minutes every morning within an hour of waking up, everyday for 4 weeks.
  Interventions: Device: Modified Dim Lamp

INTERVENTIONS:
Device: Bright Light Therapy Lamp — TRAVelite Desk Lamp manufactured by Northern Light Technologies, located in Montreal, Quebec. The light is emitted from a lamp. The florescent tubes in the box are covered with a diffusing screen to ensure even distribution of light and protection from ultraviolet light. These lamps also have a stand which enables users to place the box horizontally or vertically on most surfaces. These lamps emit light of intensity 10,000 lux.
  Arms: Bright Light Therapy Group
Device: Modified Dim Lamp — TRAVelite Desk Lamp manufactured by Northern Light Technologies, located in Montreal, Quebec. The light is emitted from a lamp. The florescent tubes in the box are covered with a diffusing screen to ensure even distribution of light and protection from ultraviolet light. These lamps also have a stand which enables users to place the box horizontally or vertically on most surfaces. These lamps have been modified to emit light of intensity 500 lux.
  Arms: Dim Light Group

SUMMARY:
Bright Light Therapy Efficacy for Depressive Symptoms Following Cardiac Surgery or Acute Coronary Syndrome: Pilot Trial (BEAM-P) is a randomized controlled trial (RCT) that seeks to assess the feasibility of conducting a full trial which would assess the efficacy of Bright Light Therapy (BLT) for improving depressive symptoms post-cardiac surgery or acute coronary syndrome.

DETAILED DESCRIPTION:
Overall Study Objective

The Bright Light Therapy Efficacy for Depressive Symptoms Following Cardiac Surgery or Acute Coronary Syndrome: Pilot Trial (BEAM-P) is a randomized controlled trial (RCT) that seeks to assess the feasibility of conducting a full trial which would assess the efficacy of Bright Light Therapy (BLT) for improving depressive symptoms post-cardiac surgery or acute coronary syndrome (ACS).

Specific Objectives

To assess the feasibility of conducting a full trial, including assessment of recruitment rate, retention rate, adherence, process time, and potential additional data values that should be measured.

Rationale

More than 50,000 Canadians undergo coronary artery bypass grafting (the most common cardiac surgery) each year and over 100,000 are hospitalized for an ACS. Of these patients, at least 15-20% experience depression. Depressed cardiac patients have a nearly 20% increased risk of all-cause mortality, increased risk of cardiac death, and increased risk of experiencing future cardiovascular events. Addressing depression and depressive symptoms in cardiac surgery and ACS patients is therefore crucial. BLT could represent a simple, safe, and cost-effective method of reducing depressive symptoms following cardiac surgery or ACS. BLT has been shown to decrease depressive symptoms in individuals with both seasonal affective disorder and non-seasonal depression in the general population, as well as in a few specific patient populations. However, the efficacy of BLT for reducing depressive symptoms post-cardiac surgery or ACS is unknown. The full BEAM Trial will be the first to study the effects of BLT in this patient population. Since BLT has not yet been investigated in cardiac patients, the feasibility of conducting a large trial of BLT in this population must be determined in order to avoid potential pitfalls and enhance the chances of success of a full trial.

Methods

We will conduct an RCT with a treatment period of 4 weeks and 12 week follow-up post-cardiac surgery or ACS. A total of 38 cardiac surgery or ACS participants will be randomized 1:1 to one of two treatment arms: 1) BLT (10,000 lux light intensity) or 2) Dim light (control group; 500 lux light intensity). Study personnel and participants will be blinded as to treatment allocation. Permutated block randomization will help ensure a balance of known and unknown confounders. Informed consent will be obtained in person from all individuals. Participants in both groups will begin using the lamps in-hospital and will continue the treatment at home for the remainder of the 4 weeks post-surgery or ACS. At baseline and day of discharge, participants will complete the Patient Health Questionnaire 9 (PHQ-9), Depression Anxiety Stress Scale short version (DASS-21), and Short Form (36) Health Survey (SF-36) questionnaires in order to determine index levels of depressive symptomology (PHQ-9, DASS-21) and health-related quality of life (SF-36). A case report form, to collect demographic and clinical information, will also be completed at baseline and day of discharge. There will be a clinic visit at week 4, when patients will return their lamp and complete questionnaires, and study personnel will complete a case report form to monitor treatment adherence. At week 12, participants will have the option to complete their questionnaires online or by mail. To compensate participants for expenses incurred due to participation (parking, childcare, opportunity costs, etc.), they will receive $25 at week 4, and a $20 prepaid VISA card after completing the questionnaires at week 12.

Significance

BLT may be a simple, cost-effective, and safe method of decreasing the severity of depression and depressive symptoms in patients following cardiac surgery or ACS. Even a small reduction in depressive symptoms could have a significant effect on the occurrence of cardiovascular events, cardiac death, and all-cause mortality in this high-risk population. The full BEAM Trial will provide regulators, health care professionals, and patients with important new information about the efficacy of BLT to decrease symptoms of depression in this population. Conducting the BEAM-P study will help ensure the success of carrying out the full BEAM Trial.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiac surgery or hospitalized for an acute coronary syndrome;
* Age ≥ 18 years;
* Score of ≥ 8 on the Patient Health Questionnaire-9;
* Able to understand and to provide informed consent in English or French; and
* Likely to be available for follow-up.

Exclusion Criteria:

* Pregnant or lactating females;
* Medical condition with a prognosis < 12 weeks;
* History of bipolar disorder, SAD, psychosis, or dementia;
* Medical condition contraindicating use of BLT (ocular or retinal pathology: glaucoma, cataracts, retinal detachment, retinopathy, diabetes);
* Medical condition that increases photosensitivity (e.g. systemic lupus erythematosus, rosacea, psoriasis, albinism);
* Current use of medication that increases photosensitivity (e.g. St John's Wort, lithium, melatonin, tetracycline, Accutane, Benzoyl peroxide, Retin-A);
* Less than one month following previous BLT;
* Light induced epilepsy or migraines; or
* Suicidal ideation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01; Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Baseline

SECONDARY OUTCOMES:
Retention rate | 12 week follow-up period
  Percentage of participants who remain in the study at week 12
Adherence rate | 4 week follow-up period
  Percentage of participants who used their lamp on ≥60% of mornings within an hour of waking for at least 25 minutes throughout the 4 week treatment period

OTHER OUTCOMES:
Determination of process time required | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Eisenberg, Principal Investigator — McGill University, Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Huffman JC, Celano CM, Beach SR, Motiwala SR, Januzzi JL. Depression and cardiac disease: epidemiology, mechanisms, and diagnosis. Cardiovasc Psychiatry Neurol. 2013;2013:695925. doi: 10.1155/2013/695925. Epub 2013 Apr 7. PMID 23653854
- [Background] Tully PJ, Baker RA. Depression, anxiety, and cardiac morbidity outcomes after coronary artery bypass surgery: a contemporary and practical review. J Geriatr Cardiol. 2012 Jun;9(2):197-208. doi: 10.3724/SP.J.1263.2011.12221. PMID 22916068
- [Background] Pincus HA, Pettit AR. The societal costs of chronic major depression. J Clin Psychiatry. 2001;62 Suppl 6:5-9. PMID 11310818
- [Background] Stewart WF, Ricci JA, Chee E, Hahn SR, Morganstein D. Cost of lost productive work time among US workers with depression. JAMA. 2003 Jun 18;289(23):3135-44. doi: 10.1001/jama.289.23.3135. PMID 12813119
- [Background] Frasure-Smith N, Lesperance F, Gravel G, Masson A, Juneau M, Talajic M, Bourassa MG. Depression and health-care costs during the first year following myocardial infarction. J Psychosom Res. 2000 Apr-May;48(4-5):471-8. doi: 10.1016/s0022-3999(99)00088-4. PMID 10880668
- [Background] Blumenthal JA. Depression and coronary heart disease: association and implications for treatment. Cleve Clin J Med. 2008 Mar;75 Suppl 2:S48-53. doi: 10.3949/ccjm.75.suppl_2.s48. PMID 18540147
- [Background] Frasure-Smith N, Lesperance F, Talajic M. Depression and 18-month prognosis after myocardial infarction. Circulation. 1995 Feb 15;91(4):999-1005. doi: 10.1161/01.cir.91.4.999. PMID 7531624
- [Background] Bush DE, Ziegelstein RC, Tayback M, Richter D, Stevens S, Zahalsky H, Fauerbach JA. Even minimal symptoms of depression increase mortality risk after acute myocardial infarction. Am J Cardiol. 2001 Aug 15;88(4):337-41. doi: 10.1016/s0002-9149(01)01675-7. PMID 11545750
- [Background] Golden RN, Gaynes BN, Ekstrom RD, Hamer RM, Jacobsen FM, Suppes T, Wisner KL, Nemeroff CB. The efficacy of light therapy in the treatment of mood disorders: a review and meta-analysis of the evidence. Am J Psychiatry. 2005 Apr;162(4):656-62. doi: 10.1176/appi.ajp.162.4.656. PMID 15800134
- [Background] Lieverse R, Van Someren EJ, Nielen MM, Uitdehaag BM, Smit JH, Hoogendijk WJ. Bright light treatment in elderly patients with nonseasonal major depressive disorder: a randomized placebo-controlled trial. Arch Gen Psychiatry. 2011 Jan;68(1):61-70. doi: 10.1001/archgenpsychiatry.2010.183. PMID 21199966
- [Background] Tuunainen A, Kripke DF, Endo T. Light therapy for non-seasonal depression. Cochrane Database Syst Rev. 2004;2004(2):CD004050. doi: 10.1002/14651858.CD004050.pub2. PMID 15106233
- [Background] Kripke DF. Light treatment for nonseasonal depression: speed, efficacy, and combined treatment. J Affect Disord. 1998 May;49(2):109-17. doi: 10.1016/s0165-0327(98)00005-6. PMID 9609674
- [Background] Niederhofer H, von Klitzing K. Bright light treatment as mono-therapy of non-seasonal depression for 28 adolescents. Int J Psychiatry Clin Pract. 2012 Sep;16(3):233-7. doi: 10.3109/13651501.2011.625123. Epub 2012 Jul 19. PMID 22809107 (Retraction: PMID 34128450 Int J Psychiatry Clin Pract. 2022 Sep;26(3):327)
- [Background] Wirz-Justice A, Bader A, Frisch U, Stieglitz RD, Alder J, Bitzer J, Hosli I, Jazbec S, Benedetti F, Terman M, Wisner KL, Riecher-Rossler A. A randomized, double-blind, placebo-controlled study of light therapy for antepartum depression. J Clin Psychiatry. 2011 Jul;72(7):986-93. doi: 10.4088/JCP.10m06188blu. Epub 2011 Apr 5. PMID 21535997
- [Background] Baxendale S, O'Sullivan J, Heaney D. Bright light therapy for symptoms of anxiety and depression in focal epilepsy: randomised controlled trial. Br J Psychiatry. 2013 May;202(5):352-6. doi: 10.1192/bjp.bp.112.122119. Epub 2013 Mar 21. PMID 23520221
- [Background] Kripke DF, Mullaney DJ, Klauber MR, Risch SC, Gillin JC. Controlled trial of bright light for nonseasonal major depressive disorders. Biol Psychiatry. 1992 Jan 15;31(2):119-34. doi: 10.1016/0006-3223(92)90199-a. PMID 1737074
- [Background] Terman M, Terman JS. Light therapy for seasonal and nonseasonal depression: efficacy, protocol, safety, and side effects. CNS Spectr. 2005 Aug;10(8):647-63; quiz 672. doi: 10.1017/s1092852900019611. PMID 16041296
- [Background] Shirani A, St Louis EK. Illuminating rationale and uses for light therapy. J Clin Sleep Med. 2009 Apr 15;5(2):155-63. PMID 19968050
- [Background] Rastad C, Ulfberg J, Lindberg P. Improvement in Fatigue, Sleepiness, and Health-Related Quality of Life with Bright Light Treatment in Persons with Seasonal Affective Disorder and Subsyndromal SAD. Depress Res Treat. 2011;2011:543906. doi: 10.1155/2011/543906. Epub 2011 Jun 13. PMID 21747994
- [Background] Reeves GM, Nijjar GV, Langenberg P, Johnson MA, Khabazghazvini B, Sleemi A, Vaswani D, Lapidus M, Manalai P, Tariq M, Acharya M, Cabassa J, Snitker S, Postolache TT. Improvement in depression scores after 1 hour of light therapy treatment in patients with seasonal affective disorder. J Nerv Ment Dis. 2012 Jan;200(1):51-5. doi: 10.1097/NMD.0b013e31823e56ca. PMID 22210362
- [Background] Naus T, Burger A, Malkoc A, Molendijk M, Haffmans J. Is there a difference in clinical efficacy of bright light therapy for different types of depression? A pilot study. J Affect Disord. 2013 Dec;151(3):1135-7. doi: 10.1016/j.jad.2013.07.017. Epub 2013 Aug 7. PMID 23972661
- [Background] Manea L, Gilbody S, McMillan D. Optimal cut-off score for diagnosing depression with the Patient Health Questionnaire (PHQ-9): a meta-analysis. CMAJ. 2012 Feb 21;184(3):E191-6. doi: 10.1503/cmaj.110829. Epub 2011 Dec 19. PMID 22184363